CLINICAL TRIAL: NCT00640874
Title: A Prospective Study to Examine the Effectiveness and Safety of Antivirals in Volunteers Who Receive Short-term Prophylaxis Against Pandemic Influenza.
Acronym: PIPET C
Status: Withdrawn | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sean Emery, Therapeutic and Vaccine Research Program, National Centre in HIV Epidemiology and Clinical Research, University of New South Wales
Other Study IDs: PIPET C
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Pandemic Influenza
Keywords: Prophylaxis; pandemic influenza; influenza A; H5N1 virus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PIPET C: Contact group members of people with diagnosed influenza who are recommended to receive NA inhibitor prophylaxis for short periods of time will be enrolled following provision of informed consent.

SUMMARY:
This aim of this project is to evaluate the efficacy of neuraminidase inhibitors as short-term prophylaxis against pandemic influenza infection in people who have close familial contact with the disease. The study is observational only. The primary measure used in this study will be the incidence of symptomatic pandemic influenza in patients receiving prophylaxis. Seroconversion to pandemic influenza, the incidence of adverse events and the relative effectiveness of oseltamivir and zanamivir prophylaxis will also be examined. This project will commence upon pandemic influenza being declared in Australia, Hong Kong or Singapore. Data will be analysed as quickly as possible to help inform the continued use of neuraminidase inhibitor therapy as a cornerstone of the public health agency response to pandemic influenza.

DETAILED DESCRIPTION:
The aim of this study is to

1. Describe the effectiveness of short-term prophylaxis against symptomatic pandemic influenza infection
2. Describe the safety of short-term prophylaxis
3. Describe the seroconversion rate against pandemic influenza among recipients of short-term prophylaxis

The study is an open label prospective cohort study. Contact group members of people with diagnosed influenza who are recommended to receive NA inhibitor prophylaxis for short periods of time will be enrolled following provision of informed consent. Each episode of short-term prophylaxis will be recorded separately.

By design it is hoped that volunteers in this study who develop symptoms and signs of pandemic influenza infection will be enrolled in the Index Case (PIPET A) protocol with follow-up as required.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Intention to commence or have commenced short-term prophylaxis with a neuraminidase inhibitor in individuals who have been exposed to the pandemic virus

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Contact group members of people with diagnosed influenza who are recommended to receive NA inhibitor prophylaxis for short periods of time will be enrolled following provision of informed consent. Each episode of short-term prophylaxis will be recorded separately.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The primary measure used in this study will be the incidence of symptomatic pandemic influenza in patients receiving prophylaxis. | One month

SECONDARY OUTCOMES:
Seroconversion to pandemic influenza, the incidence of adverse events and the relative effectiveness of oseltamivir and zanamivir prophylaxis will also be examined. | One month

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Dwyer, Principal Investigator — Westmead Hospital
Locations (8):
- Australia (8):
  - St Vincent's Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Westmead Hospital, Sydney, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia